CLINICAL TRIAL: NCT00827554
Title: A Clinical Randomized Control Trial of Combination TACE With and Without Low-molecular-weight Heparin in Hepatocellular Carcinoma
Brief Title: The Role of Low Molecular Weight Heparins in Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-011
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver Neoplasms; Liver Diseases; Digestive System Diseases; Digestive System Neoplasms; Carcinoma, Hepatocellular; Gastrointestinal Neoplasms; Adenocarcinoma; Hepatocellular carcinoma; Neoplasms; Transarterial chemoembolization; Nadroparin; low-molecular-weight heparin; chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Liver Diseases; Digestive System Diseases; Digestive System Neoplasms; Gastrointestinal Neoplasms; Adenocarcinoma; Neoplasms | interventions — Heparin, Low-Molecular-Weight; Nadroparin; halofantrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMWH plus TACE (Experimental): 50 HCC patients will be allocated to receive Nadroparin 4100 AXa iu twice daily 3 days after TACE which lasted for 6 weeks
  Interventions: Drug: LMWH; Procedure: TACE
- TACE alone (Active Comparator): 50 HCC patients randomly assigned to receive TACE without LMWH
  Interventions: Drug: LMWH; Procedure: TACE

INTERVENTIONS:
Drug: LMWH — Nadroparin Ca 4100 AXa iu twice daily lasted for 6 weeks
  Other Names: fraxiparine; GlaxoSmithKline
Procedure: TACE — transarterial chemoembolization with lipiodol 1-1.5ml/cm tumor diametres，pharmorubicin 20mg，5-Fu 1g and Carboplatin 150mg。
  Other Names: transarterial embolization/chemoembolization

SUMMARY:
Hepatocellular carcinoma (HCC) is a major tumor type worldwide, especially in China as the sequence of hepatitis B and liver cirrhosis. Activation of the coagulation system occurs commonly in patients with malignancy. Several studies have suggested that anticoagulant therapy may improve survival in patients with malignancy. The low molecular weight heparins (LMWHs) lend themselves to such studies because of their effects in experimental models of malignancy and the relative ease of administration compared with unfractionated heparin. The purpose of the present RCT was to determine whether addition of LMWH to transarterial chemoembolization (TACE) would improve HCC patient outcome compared with TACE alone.

DETAILED DESCRIPTION:
100 patients will be randomly assigned to receive either TACE alone or TACE plus LMWH. A block of every 4 participants and a stratified randomization according to portal vein cancer emboli will be used to restrict randomization. LMWH consisted of nadroparin Ca will be given at a dose of 4100 U twice daily during 6 weeks after TACE. The time to progression(TTP) and overall survival within two years will be used to evaluate the effect of LMWH on HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Adults patients with a diagnosis of HCC which is not amenable to surgical resection, liver transplantation or local ablative therapy
2. Without metastasis out of liver
3. Patients must have at least one tumor lesion that meets both of the following criteria:

   1. The lesion can be accurately measured in at least one dimension according to RECIST criteria
   2. The lesion has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
4. ECOG performance status (PS) <2
5. No prior targeted antiangiogenic therapy. Metronomic chemotherapies are allowed. At least 4 weeks since prior systemic chemotherapy
6. Child-Pugh class A or B
7. No significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis
8. Ability to understand the protocol and to agree to and sign a written informed consent document -

Exclusion Criteria:

1. HBSAg(-)，AFP(-).
2. prothrombin time prolonged more than 4s.
3. blood platelets count less than 50000/L.
4. Renal failure requiring dialysis.
5. Child-Pugh class C hepatic impairment.
6. clinically significant gastrointestinal bleeding within 30 days prior to study entry.
7. History of organ allograft.
8. Substance abuse (current), psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
9. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
10. Pregnant or breast-feeding patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
time-to-progression(TTP) | 1 year

SECONDARY OUTCOMES:
The overall response rate | 1 year
Overall survival (OS) | 1 year
bleeding complication rate | 6 weeks
Progression Free Survival (PFS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China